CLINICAL TRIAL: NCT07327983
Title: Topical 20% Azelaic Acid Versus 4% Hydroquinone in Epidermal Melasma: A Randomized Controlled Trial
Brief Title: Azelaic Acid 20% vs Hydroquinone 4% in Epidermal Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gujranwala medical college District Headquarters Hospital, Gujranwala (Other)
Responsible Party: Principal Investigator, Yasan Saaqib, 5th year resident, Gujranwala medical college District Headquarters Hospital, Gujranwala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB.23/GMC
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Melasma; Melasma (Facial Melasma)
Keywords: Melasma; Azelaic Acid; Hydroquinone; Topical Therapy; Hyperpigmentation; Comparative Study; Dermatology
MeSH Terms: conditions — Melanosis; Hyperpigmentation | interventions — azelaic acid

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to receive either topical 20% azelaic acid or topical 4% hydroquinone for 12 weeks.
Who Masked: Participant
Masking Description: Participants were blinded to treatment allocation. Treating clinicians and study staff were aware of group assignments. The statistician analyzing the data received coded datasets and was blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GroupA (Experimental): Subjects were randomised into two intervention groups of 73 each by paralel assignment .
  Group A (Azelaic Acid 20%) Description Group A Participants were assigned to 20%Azalic acid daily application for 12weeks as intervention for treatment of Melasma.
  Interventions: Drug: Topical Azelaic Acid 20% Cream
- GroupB (Active Comparator): Group B (Hydroquinone 4%) Description the other grouphad also 73 participants.They were assigned to 4%Hydroquinone daily application for 12 as intervention for treatment of Melasma.
  Interventions: Drug: Topical 4% hydroquinone cream

INTERVENTIONS:
Drug: Topical Azelaic Acid 20% Cream — Topical azelaic acid 20% cream was applied in intervention group to affected facial areas once daily for 12 weeks. The intervention is used to reduce hyperpigmentation in patients with melasma.
  Arms: GroupA
Drug: Topical 4% hydroquinone cream — The other intervention isTopical application of hydroquinone 4% cream to affected facial areas once daily for 12 weeks.
  Arms: GroupB

SUMMARY:
Melasma is a common skin condition that causes dark patches on the face and can significantly affect quality of life. This study compared two commonly used topical treatments, 20% azelaic acid and 4% hydroquinone, in adults with epidermal melasma.

Participants with epidermal melasma were randomly assigned to receive either azelaic acid 20% or hydroquinone 4% for a period of 12 weeks. The severity of melasma was assessed at baseline and monthly using the Melasma Area and Severity Index (MASI) score. Side effects such as irritation, redness, burning, itching, and dryness were also monitored throughout the study.

The purpose of this study was to compare the effectiveness and safety of azelaic acid and hydroquinone in reducing melasma severity and to determine whether azelaic acid can be used as a safe alternative to hydroquinone.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted in the Dermatology Department of Gujranwala Medical College Hospital, Gujranwala, from 4 May 2025 to 3 August 2025. The study was designed to compare the efficacy and safety of topical 20% azelaic acid and 4% hydroquinone in the treatment of epidermal melasma.

A total of 146 patients with clinically diagnosed epidermal melasma confirmed by Wood's lamp examination were enrolled. Patients of any age and gender were eligible. Exclusion criteria included dermal or mixed-type melasma, active skin infections, history of keloid formation, recent use of other depigmenting agents, photosensitive disorders, pregnancy or lactation, and refusal to provide written informed consent.

After obtaining informed consent, participants were randomly assigned to one of two treatment groups in a parallel design. Group A received topical azelaic acid 20%, and Group B received topical hydroquinone 4%. Participants were blinded to their treatment allocation, while treating clinicians and research staff were aware of the assigned treatment. The statistician analyzing the data was blinded to group allocation.

Both treatments were administered for a duration of 12 weeks. Participants were evaluated at baseline and then monthly. All participants were advised to use broad-spectrum sunscreen throughout the study period. Treatment compliance and adverse effects were assessed at each follow-up visit. Any adverse effects such as erythema, burning, itching, or dryness were managed with supportive care, including emollients or antihistamines if required.

The primary outcome measure was treatment efficacy, assessed by the change in Melasma Area and Severity Index (MASI) score from baseline to the end of the 12-week treatment period. Secondary outcomes included the rate of improvement over time and the safety and tolerability of both treatments.

MASI scoring was performed using a standardized method that evaluates the area of involvement, darkness, and homogeneity of melasma across four facial regions: forehead, right malar region, left malar region, and chin. Clinical photographs were also obtained to support clinical assessment.

Data were analyzed using statistical software. Quantitative variables were summarized as means and standard deviations, and qualitative variables as frequencies and percentages. Between-group comparisons of MASI scores were performed using independent-samples t-tests, with a p-value of less than 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed epidermal melasma confirmed by Wood's lamp examination
* Male or female participants of any age
* Willingness to provide written informed consent
* Ability to comply with study procedures and follow-up visits

Exclusion Criteria:- Dermal or mixed-type melasma

* Active cutaneous or facial skin infection
* History of keloid formation
* Recent use of other topical or systemic depigmenting agents
* Presence of photosensitive disorders
* Pregnancy or lactation
* Refusal or inability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2025-05-04 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Change in Melasma Area and Severity Index (MASI) Score | Baseline to 12 weeks
  The primary outcome was treatment efficacy, assessed by the change in the Melasma Area and Severity Index (MASI) score from baseline to the end of the 12-week treatment period. MASI evaluates the severity of melasma based on area of involvement, darkness, and homogeneity across four facial regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Gujranwala Medical College Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
We will do it after publication